CLINICAL TRIAL: NCT04921306
Title: Targeting the Beta-2-adrenergic Pathway to Improve Skeletal Muscle Glucose Uptake in Obese Humans
Brief Title: Obese Human Beta-2-adrenergic Stimulation and Muscle Glucose Uptake
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: Eurostars (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NL76746.068.21
Record Dates: First submitted 2021-05-25; First posted 2021-06-10 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clenbuterol hydrochloride (Experimental): Subjects will ingest clenbuterol hydrochloride capsules (20 microgram/each) twice daily (40 microgram/day) for a maximum of 28 days.
  Subjects that received the clenbuterol hydrochloride capsules (at random) in the first study period will receive the placebo capsules during the second study period.
  Interventions: Drug: Clenbuterol Hydrochloride
- Placebo (Placebo Comparator): Subjects will ingest placebo capsules matching the clenbuterol hydrochloride capsules one time per day for a maximum of 28 days.
  Subjects that received the placebo capsules (at random) in the first study period will receive the clenbuterol hydrochloride capsules during the second study period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clenbuterol Hydrochloride — Daily ingestion of clenbuterol hydrochloride capsules (40 microgram/day) for a total period of 28 days with a wash-out period of at least 6-8 weeks.
  Arms: Clenbuterol hydrochloride
Drug: Placebo — Daily ingestion of placebo capsules for a total period of 28 days with a wash-out period of at least 6-8 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of four weeks clenbuterol/placebo supplementation on skeletal muscle glucose disposal in overweight/obese male and (postmenopausal) female volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian;
2. Male or (postmenopausal; defined as 1 year after the last cycle) female;
3. Age between 40-70 years;
4. BMI: 27-35 kg/m2;

Exclusion Criteria:

1. Not meeting all inclusion criteria
2. Cardiovascular disease (determined by means of questionnaires, heart rate/blood pressure measurements and an ECG)
3. Respiratory diseases (including asthma, bronchitis and COPD);
4. Unstable body weight (weight gain or loss > 3 kg in the last three months);
5. Intention to lose or gain body weight (e.g. with caloric restriction or physical activity)
6. Excessive alcohol and/or drug abuse;
7. Hypokalaemia;
8. Hyperthyroidism
9. Anaemia;
10. Epilepsy;
11. Smoking;
12. Renal and/or liver insufficiency;
13. Diagnosed with type 1 or type 2 diabetes mellitus;
14. Any contra-indications to MRI scanning. These contra-indications include patients with:

    1. Electronic implants such as pacemakers, defibrillators or neurostimulators
    2. Central nervous system aneurysm clip
    3. Some hearing aids (such as cochlear implant) and artificial (heart) valves which are contraindicated for MRI/MRS
    4. Iron containing corpora aliena in the eye or brains
    5. Claustrophobia
15. Participation in another biomedical study within 1 month before the first study visit, possibly interfering with the study results;
16. Medication use known to hamper subject's safety during the study procedures;
17. Subjects who do not want to be informed about unexpected medical findings;
18. Subjects who do not want that their treating physician to be informed;
19. Inability to participate and/or complete the required measurements;
20. Participation in organised or structured physical exercise (>2h per week);
21. Any condition, disease or abnormal laboratory test result that, in the opinion of the Investigator, would interfere with the study outcome, affect trial participation or put the subject at undue risk;

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
insulin-stimulated fluorodeoxyglucose (18F-FDG) uptake in quadriceps muscle. | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on insulin-stimulated 18F-FDG uptake in quadriceps muscle as assessed using radio-active labelled tracer (18F-FDG) in positron emission tomogaphy magnetic resonance imaging (PET-MRI).

SECONDARY OUTCOMES:
insulin-stimulated 18F-FDG uptake in BAT | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on insulin-stimulated 18F-FDG uptake in BAT as assessed using radio-active labelled tracer (18F-FDG) in PET-MRI.

OTHER OUTCOMES:
Body weight | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on body weight
Lean mass | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on lean mass as assessed by Bodpod measurement
Fat mass | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on fat mass as assessed by Bodpod measurement
Glucose infusion rate (GIR) | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on glucose-infusion rate (GIR) during a one-step hyperinsulinemic-euglycemic clamp
Plasma insulin concentrations | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on plasma insulin concentrations
Plasma glucose concentrations | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on plasma glucose concentrations
Plasma free fatty acid (FFA) concentrations | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on plasma FFA concentrations
Plasma triacylglycerol (TAG) concentrations | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on plasma (TAG) concentrations
Heart rate | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on heart rate as assessed by means of an automated cuff
Blood pressure | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on blood pressure (systolic and diastolic blood pressure) as assessed by means of an automated cuff
Energy expenditure | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on energy expenditure as measured by indirect calorimetry
Substrate oxidation | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on substrate oxidation as measured by indirect calorimetry
Sleeping energy expenditure | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on sleeping energy expenditure as assessed by means of whole-room indirect calorimetry
Substrate oxidation during sleep | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on substrate oxidation during sleep as assessed by means of whole-room indirect calorimetry
Skeletal muscle gene expression | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on skeletal muscle gene expression of insulin signalling and beta-adrenergic pathways as determined in muscle biopsies by means of RT-qPCR
Skeletal muscle protein expression | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on skeletal muscle protein expression of insulin signalling and adrenergic signalling pathways as determined in muscle biopsies by means of Western blot
Femoral artery flow mediated dilation | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on FMD as assessed by means of echo-doppler
skeletal muscle GLUT4 translocation | 4 weeks
  Comparison between prolonged (4 weeks) clenbuterol hydrochloride or placebo supplementation on skeletal muscle GLUT4 translocation as assessed by means of wide-field microscopy in skeletal muscle biopsies

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Netherlands